CLINICAL TRIAL: NCT04297982
Title: The Effect of Mandala Activity on Psychological Symptoms, Anxiety and Depression Level of Adolescents Receiving Cancer Treatment
Brief Title: Mandala Activity and Adolescents With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Meltem Gürcan, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AkUn
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Nursing
Keywords: cancer; adolescent; mandala; anxiety; depression
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Mandala activity) (Experimental): Scales were applied to the experimental group in the first encounter with the adolescent (pre-test). Then, a total of two sessions of individual mandala activities were performed at least 48 hours apart. Each adolescent freely drawn and painted the unstructured mandala on white paper, starting from the center and expanding. The same scales were reapplied last (post-test).
  Interventions: Other: Mandala Activity; Other: Routine nursing care
- Control group (Other): Scales were applied to the control group with an interval of 5 days and received routine nursing care (pre-test, post-test).
  Interventions: Other: Routine nursing care

INTERVENTIONS:
Other: Mandala Activity — Mandala is a method of expressing one's feelings and thoughts. The person draws and paints the paper in a round shape.
  Arms: Intervention group (Mandala activity)
Other: Routine nursing care — Interventions routinely implemented by nurses in the clinic

SUMMARY:
Aim: The aim of this study is to determine the effect of mandala activity on adolescents receiving cancer treatment on psychological symptoms and anxiety/depression level.

Method: The study was conducted as a randomized controlled experimental study with adolescents aged 12-17 years receiving cancer treatment in Akdeniz University Hospital Pediatric Hematology and Oncology Clinic. The sample group was composed of 30 adolescents in the experimental group and 30 adolescents in the control group using the closed envelope system in accordance with the selection criteria of the sample. The experimental group was given 2 sessions of mandala drawing and staining activity with music at least 48 hours apart. In the study, individual activity was preferred. In each session, adolescents were allowed to draw and stain a mandala. 'Data Collection Form' before the first session, 'Memorial Symptom Assessment Scale', ''Hospital Anxiety and Depression Scale were applied to the experimental group before and after the first session. The same data collection tools were applied to the control group at 48 hours intervals without any activity.

DETAILED DESCRIPTION:
Type of the Study This research; This is a randomized controlled experimental study to determine whether mandala activity applied to adolescents receiving cancer treatment has an effect on psychological symptoms and anxiety / depression level.

Place and Time of the Study The research was carried out in Antalya Akdeniz University Hospital, Child Hematology / Oncology Clinic. The research data were collected by the researcher between March 2019 and February 2020. Akdeniz University Child Hematology and Oncology Clinic is a 32-bed institution where children between 0-18 years old receive inpatient treatment and care. It is forbidden to visit the clinic to protect patients from infection, thereby providing a calm environment in the clinic. The rooms are double and single.

Mandala activity at a normal room temperature (average 25 ° C), in terms of being bright enough and a comfortable environment for adolescents; It was planned to have a room that was spacious, clean, with a window opening (not opening to the corridor) and in sunlight, and it was decided that the most suitable environment in the clinic was the patient's own room.

Sample of the Research The sampling of the study was composed of all adolescents who received cancer treatment in Akdeniz University Hospital Child Hematology / Oncology Clinic. Adolescents who accepted to participate in the study on a voluntary basis and having the inclusion criteria constituted the sample of the study. The sample group was formed in accordance with the sample selection criteria and divided into two as experimental and control groups. As a result of the power analysis, the sample group with 80% power and 0.05 error margin; The experimental group 30 and the control group 30 were planned to form a total of 60 children receiving cancer treatment.

Data Collection Tools In this study; Two scales were used for the descriptive features of the Personal Information Form, Memorial Symptom Evaluation Scale Psychological Sub-Dimension (MSDÖ-P) and Hospital Anxiety and Depression Scale (Adolescent Age Group Form).

Prior to the research, permission was obtained from the Antalya Akdeniz University Clinical Research Ethics Committee regarding the method and design of the study (Decision No: 492, Date: 11.07.2018). After obtaining the approval of the ethics committee, necessary verbal and written permissions were obtained from Akdeniz University Hospital. Permission was obtained to use the Memorial Symptom Assessment Scale, which was adapted to Turkish for children aged 10-18 by Atay in 2008, validity and reliability study. Permission was obtained via e-mail to use the Hospital Anxiety and Depression Scale, which was validated for validity and reliability in the adolescent age group by Erkan in 2014.

Before starting the study, it was explained to the adolescent about the purpose, duration, fee of the research, all information will be kept confidential and will not be used anywhere other than the thesis. In addition, informed consent was obtained from the adolescent by explaining that there will be no difficulty in participating in the study and that the study is based on volunteering, and that they can leave whenever they want during the application phase. Before the application of the research, the parent was informed about the research in written or verbally. The researcher attended mandala education before the thesis study.

Mandala Activity (İnterventation Group) Scales were applied to the experimental group in the first encounter with the adolescent (pre-test). One day later, one session of individual mandala activity were performed. Later at least 48 hours, also one session of individual mandala activity. Each adolescent created two seans mandala and freely drawn and painted the unstructured mandala on white paper, starting from the center and expanding. A day after the second session mandala activity the same scales were reapplied last (post-test).

Control Group Scales were applied to the control group with an interval of 5 days and received routine nursing care (pre-test, post-test).

Mandala Activity Application Steps

* Researchers ensured that the patient is not in times such as sleep or meal time.
* The best time for the activity was determined by exchanging ideas with the patient.
* Hygienic rules were taken care of (Washing hands and wiping the materials with alcohol cotton).
* A comfortable environment has been provided for activities (the room is bright enough, closing the room door to prevent noise, lifting the back of the bed with the patient in a sitting position, and adjusting the height of the table brought in front of the patient).
* Sample videos on how to draw mandala were watched before the application.
* Adolescents were told that the beauty of the drawings was not important, as the mandala is a means of expression and sharing.
* In the individual mandala activity, the drawings were made with classical / instrumental music.
* It was provided to paint and then paint before painting from the center on the picture paper without disturbing the order.
* When created mandala, all the drawings and paintings were made inside the circles drawn together.
* Adolescents are free to choose colors and shapes during the individual mandala activity.
* Unless the adolescents asked for help, the researcher did not intervene in the mandala drawing

ELIGIBILITY:
Inclusion Criteria:

* Must be able to read and speak Turkish
* Clinical diagnosis of cancer disease
* The ages of 12-17.
* The duration of diagnosis is at least 2 months
* Must be have cancer treatment,

Exclusion Criteria:

* The patient is in the terminal period

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Memorial Symptom Assessment Scale Psychological Sub Dimension | 5 day
  Memorial Symptom Assessment Scale is a scale developed by Portenoy et al. In 1994 in order to determine the symptoms experienced by patients with cancer diagnosis in the last week. In 2000, Collins et al. Adapted the scale to adults by carrying out the validity and reliability study of children aged 10-18 years of age. Adaptation, validity and reliability studies were carried out in 2007 by Atay et al. The psychological sub-dimension of the scale was used in the planned study. In this study, Cronbach's alpha value of all items of the scale was determined as .90. The statistically significant increase in the mean score of psychological symptoms in posttest measurement in the intervention group is the success criterion of the study. Significance level is set at p<0.05 in analyzes. No statistically significant difference is expected in the pretest posttest mean scores of the control group.
Hospital Anxiety and Depression Scale | 5 day
  Hospital Anxiety and Depression Scale was developed in 1983 by Zigmond and Snaith. The Turkish version of the scale in the adult age group was made in 1997 by Aydemir et al. The application time of the scale is 2-5 minutes. In 2014, Erkan adapted to Turkish culture and language in the 12-17 adolescent age group, and its validity and reliability study was performed. The scale consists of 14 items, it includes the 7-item Anxiety subscale and Depression subscale. In each item, a score of 0-3 is obtained by choosing one of the four-likert type options.
  The statistically significant increase in the mean score of anxiety and depression in posttest measurement in the intervention group is the success criterion of the study. Significance level is set at p<0.05 in analyzes. No statistically significant difference is expected in the pretest posttest mean scores of the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Sevcan ATAY TURAN, PhD, Study Director — Akdeniz University
Locations (1):
- Meltem Gürcan, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malchiodi, C. A. Medical art therapy with children: Jessica Kingsley Publishers; 1999,
- [Background] Portenoy RK, Thaler HT, Kornblith AB, Lepore JM, Friedlander-Klar H, Kiyasu E, Sobel K, Coyle N, Kemeny N, Norton L, et al. The Memorial Symptom Assessment Scale: an instrument for the evaluation of symptom prevalence, characteristics and distress. Eur J Cancer. 1994;30A(9):1326-36. doi: 10.1016/0959-8049(94)90182-1. PMID 7999421
- [Background] Kim, S.-i., Ghil, J.-H., Choi, E.-Y., Kwon, O.-S., & Kong, M. A computer system using a structured mandala to differentiate and identify psychological disorders. The Arts in Psychotherapy. 2014; 41 (2): 181-186.
- [Background] Kostyunina, N. Y., & Drozdikova-Zaripova, A. R. Adolescents' school anxiety correction by means of mandala art therapy. International Journal of Environmental and Science Education. 2016; 11 (6): 1105-1116.
- [Background] Wagner, H. The use of music and mandala to explore the client/therapist relationship in a therapeutic day school. Qualitative Inquiries in Music Therapy. 2012; 7.
- [Background] Stinley, N. E., Norris, D. O., & Hinds, P. S. Creating mandalas for the management of acute pain symptoms in pediatric patients. Art Therapy. 2015; 32 (2): 46-53.
- [Background] Serokowa D, Kreska B. [Rabies]. Przegl Epidemiol. 1975;29(1):117-20. No abstract available. Polish. PMID 1118635
- [Derived] Gurcan M, Atay Turan S. The effectiveness of mandala drawing in reducing psychological symptoms, anxiety and depression in hospitalised adolescents with cancer: A randomised controlled trial. Eur J Cancer Care (Engl). 2021 Nov;30(6):e13491. doi: 10.1111/ecc.13491. Epub 2021 Jul 29. PMID 34322921